CLINICAL TRIAL: NCT05139017
Title: A Phase 2/3 Multicenter, Open-label, Randomized, Active-Control Study of Zilovertamab Vedotin (MK-2140) in Combination With Standard of Care in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (waveLINE-003)
Brief Title: A Study of Zilovertamab Vedotin (MK-2140) in Combination With Standard of Care in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (rrDLBCL) (MK-2140-003)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2140-003; VLS-101 (Other: Velos Bio); MK-2140-003 (Other: MSD); waveLINE-003 (Other: MSD); 2022-502646-27-00 (Registry Identifier: EU CT); U1111-1285-0898 (Registry Identifier: UTN)
Record Dates: First submitted 2021-11-11; First posted 2021-12-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: DLBCL; Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Gemcitabine; Oxaliplatin; Bendamustine Hydrochloride; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: In Part 1, Dose Confirmation will be determined by modified toxicity probability interval (mTPI) design, where participants will be assigned to two treatment groups, cohort: A (zilovertamab vedotin in combinatio with R-GemOx) in parallel with cohort B (zilovertamab vedotin in combination with BR). Part 2 will be an Efficacy Expansion (cohorts A & B) where all participants in each cohort will be assigned to 2 treatment groups for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ZV + R-GemOx (Part 1) (Experimental): Participants in this arm will receive doses of ZV (from 1.5 mg/Kg up to 2.5 mg/Kg) plus Rituximab 375 mg/m^2, Gemcitabine 1000 mg/m^2 and Oxaliplatin 100 mg/m^2 (R-GemOx) given intravenously on Day 1 of repeated 21-day cycles. Treatment will continue for up to 6 cycles.
  Interventions: Biological: Zilovertamab vedotin; Biological: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Granulocyte Colony-Stimulating Factor (G-CSF)
- ZV + R-GemOx (Part 2) (Experimental): Using the recommended Phase 2 dose (RP2D) dose of ZV plus R-GemOx from Part 1, participants will receive ZV plus R-GemOx given intravenously on Day 1 of repeated 21-day cycles. Treatment will continue for up to 6 cycles or until progressive disease or discontinuation.
  Interventions: Biological: Zilovertamab vedotin; Biological: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Granulocyte Colony-Stimulating Factor (G-CSF)
- R-GemOx (active control for Part 2) (Active Comparator): Participants will receive R-GemOx given intravenously on Day 1 of repeated 21-day cycles. Treatment will continue for up to 6 cycles or until progressive disease or discontinuation.
  Interventions: Biological: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin
- ZV + BR (Part 2) (Experimental): Using RP2D from Part 1, participants will receive ZV plus Rituximab 375 mg/m^2, given intravenously on Day 1 and Bendamustine 90 mg/m^2 given intravenously on Day 1 and 2, of repeated 21-day cycles. Treatment will continue for up to 6 cycles or until progressive disease or discontinuation.
  Interventions: Biological: Zilovertamab vedotin; Biological: Rituximab; Drug: Bendamustine; Drug: Granulocyte Colony-Stimulating Factor (G-CSF)
- Bendamustine Rituximab (BR) (Active Comparator): Participants will receive Rituximab 375 mg/m^2, given intravenously on Day 1 Bendamustine 90 mg/m^2 given intravenously on Day 1 and 2 of repeated 21-day cycles. Treatment will continue for up to 6 cycles or until progressive disease or discontinuation.
  Interventions: Biological: Rituximab; Drug: Bendamustine
- ZV + BR (Part 1) (Experimental): Participants in this arm will receive doses of ZV (from 1.5 mg/Kg up to 2.5 mg/Kg) plus Rituximab 375 mg/m^2, Bendamustine 90 mg/m^2 (BR) given intravenously on Day 1 and 2 of repeated 21-day cycles. Treatment will continue for up to 6 cycles.
  Interventions: Biological: Zilovertamab vedotin; Biological: Rituximab; Drug: Bendamustine; Drug: Granulocyte Colony-Stimulating Factor (G-CSF)

INTERVENTIONS:
Biological: Zilovertamab vedotin — Intravenous (IV) Infusion 1.5 mg/kg, 1.75 mg/kg, 2.0 mg/kg, 2.25 mg/kg, 2.5 mg/kg
  Other Names: MK-2140; VLS-101
  Arms: ZV + BR (Part 1); ZV + BR (Part 2); ZV + R-GemOx (Part 1); ZV + R-GemOx (Part 2)
Biological: Rituximab — IV Infusion 375 mg/m^2
  Other Names: Rituxan®/mabthera; Truxima® (rituximab-abbs); RUXIENCE®, RIABNI®
Drug: Gemcitabine — IV Infusion 1000 mg/m^2
  Other Names: Gemzar®
  Arms: R-GemOx (active control for Part 2); ZV + R-GemOx (Part 1); ZV + R-GemOx (Part 2)
Drug: Oxaliplatin — IV Infusion 100 mg/m^2
  Other Names: Eloxatin®
  Arms: R-GemOx (active control for Part 2); ZV + R-GemOx (Part 1); ZV + R-GemOx (Part 2)
Drug: Bendamustine — IV Infusion 90 mg/m^2
  Other Names: Bendeka®; Treanda®; Belrapzo®
  Arms: Bendamustine Rituximab (BR); ZV + BR (Part 1); ZV + BR (Part 2)
Drug: Granulocyte Colony-Stimulating Factor (G-CSF) — Prophylactic G-CSF will be administered at each cycle of zilovertamab vedotin as per the institutional guidelines.
  Arms: ZV + BR (Part 1); ZV + BR (Part 2); ZV + R-GemOx (Part 1); ZV + R-GemOx (Part 2)

SUMMARY:
The purpose of this Phase 2/3, randomized, multisite, open-label, dose confirmation, and expansion study is to evaluate the safety, and efficacy of zilovertamab vedotin (ZV) in combination with standard of care options for the treatment of rrDLBCL. This study will be divided into 2 parts: Dose Confirmation (Part 1) and Efficacy Expansion (Part 2) and will enroll participants who are at least 18 years of age with rrDLBCL. The hypotheses are: ZV in combination with rituximab, gemcitabine, and oxaliplatin (R-GemOx) is superior to R-GemOx with respect to progression-free survival (PFS) per Lugano response criteria by blinded independent review committee (BICR); and that ZV in combination with bendamustine rituximab (BR) is superior to BR with respect to PFS per Lugano response criteria by BICR.

With protocol amendment 4 (effective: 04-April-2024), enrollment in Cohort B (study arms Bendamustine Rituximab [BR] and ZV + BR) is discontinued. No efficacy outcome analysis and hypothesis testing will be conducted for Cohort B.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed diagnosis of Diffuse Large B-Cell Lymphoma (DLBCL).
* Has radiographically measurable DLBCL per the Lugano Response Criteria, as assessed locally by the investigator.
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2 within 7 days prior to study treatment initiation.
* Has adequate organ function.
* Is able to provide new or archival tumor tissue sample not previously irradiated.

Zilovertamab vedotin plus R-GemOx, or R-GemOx study arms:

* Has relapsed or refractory DLBCL and is ineligible for or have failed autologous stem-cell transplant (ASCT) and have failed at least 1 line of prior therapy.
* Has post-chimeric antigen receptor T (post-CAR-T) cell therapy failure or is ineligible for CAR-T cell therapy.

Not applicable with protocol amendment 4: Zilovertamab vedotin plus Bendamustine Rituximab (BR), and Bendamustine Rituximab study arms:

* Has relapsed or refractory DLBCL and is ineligible for or have failed ASCT and have failed at least 2 lines of prior therapy.
* Has post-CAR-T therapy failure or is ineligible for CAR-T cell therapy.

Exclusion Criteria:

* Not applicable with protocol amendment 4: Has history of transformation of indolent disease to DLBCL
* Has received solid organ transplant at any time.
* Has received a diagnosis of primary mediastinal B-cell lymphoma (PMBCL).
* Has clinically significant (ie, active) cardiovascular disease or serious cardiac arrhythmia requiring medication.
* Has ongoing graft-versus-host disease (GVHD) of any grade, or is receiving treatment for their GVHD.
* Has clinically significant pericardial or pleural effusion.
* Has ongoing Grade >1 peripheral neuropathy.
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
* Has a demyelinating form of Charcot-Marie-Tooth disease.
* Has contraindication to any of the study intervention components including but not limited to prior anaphylactic reaction.
* Has received prior systemic anticancer therapy, including investigational agents within 4 weeks prior to the first dose of study intervention.
* Has received prior radiotherapy within 4 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Has ongoing corticosteroid therapy.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention.
* Has known active central nervous system (CNS) lymphoma involvement or active CNS involvement by lymphoma. Participants with prior CNS involvement are eligible if their CNS disease is in radiographic, cytological (for cerebrospinal fluid disease), and clinical remission.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known active Hepatitis C virus infection.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2027-09-24 (Estimated); Study Completion 2027-09-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experienced dose-limiting toxicities (DLTs) in Part 1 | Up to ~6 weeks
  The CTCAE, Version 5.0 will be used to grade the severity of AEs in this study. DLTs will be reported for Part 1 of this study.
Number of participants who experienced an adverse event (AE) | Up to ~68 months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who experienced an AE will be reported.
Number of participants who discontinued study treatment due to an AE | Up to ~68months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who discontinued study treatment due to an AE will be reported.
Overall survival (OS) | Up to ~35 months
  OS, defined as the time from randomization to death due to any cause will be reported.
Progression-free survival (PFS) | Up to ~26 months
  PFS, defined as the time from randomization to the first documented disease progression per Lugano response criteria as assessed by BICR or death due to any cause, whichever occurs first will be presented.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to ~26 months
  ORR, defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) per Lugano criteria as assessed by BICR will be presented.
Duration of response (DOR) | Up to ~26 months
  DOR, defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first, will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (113):
- United States (18):
  - Palo Verde Hematology/ Oncology Center, Ltd. ( Site 0175), Glendale, Arizona
  - Bass Medical Group ( Site 0166), Walnut Creek, California
  - Innovative Clinical Research Institute ( Site 0122), Whittier, California
  - Boca Raton Regional Hospital- Lynn Cancer Institute ( Site 0163), Boca Raton, Florida
  - Clermont Oncology Center ( Site 0174), Clermont, Florida
  - Saint Elizabeth Medical Center Edgewood ( Site 0165), Edgewood, Kentucky
  - University of Kentucky Chandler Medical Center ( Site 0158), Lexington, Kentucky
  - Norton Women's and Children's Hospital-Norton Cancer Institute - St. Matthews ( Site 0133), Louisville, Kentucky
  - University of Maryland ( Site 0123), Baltimore, Maryland
  - Dana-Farber Cancer Institute-Lymphoma ( Site 0111), Boston, Massachusetts
  - University of Massachusetts Medical School ( Site 0119), Worcester, Massachusetts
  - Corewell Health ( Site 0162), Grand Rapids, Michigan
  - St. Vincent Frontier Cancer Center-Research ( Site 0108), Billings, Montana
  - Comprehensive Cancer Centers of Nevada ( Site 0168), Las Vegas, Nevada
  - Atlantic Health System ( Site 0116), Morristown, New Jersey
  - New York Medical College ( Site 0113), Valhalla, New York
  - Vanderbilt University Medical Center-Vanderbilt-Ingram Cancer Center ( Site 0156), Nashville, Tennessee
  - Blue Ridge Cancer Care ( Site 0169), Roanoke, Virginia
- Argentina (5):
  - Hospital Italiano de Buenos Aires ( Site 2203), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 2205), Mar del Plata, Buenos Aires
  - Hospital Aleman ( Site 2200), Buenos Aites, Buenos Aires F.D.
  - Hospital Privado Universitario de Córdoba ( Site 2202), Córdoba, Córdoba Province
  - Instituto Alexander Fleming ( Site 2201), CABA
- Australia (3):
  - Townsville University Hospital ( Site 1800), Douglas, Queensland
  - Grampians Health ( Site 1802), Ballarat, Victoria
  - Royal Perth Hospital-Haematology ( Site 1801), Perth, Western Australia
- Brazil (4):
  - Hospital Erasto Gaertner ( Site 2302), Curitiba, Paraná
  - Liga Norte Riograndense Contra o Câncer ( Site 2305), Natal, Rio Grande do Norte
  - Hospital Paulistano ( Site 2300), São Paulo
  - Pesquisa Clínica do Serviço de Hematologia do Hospital das Clínicas da FMUSP ( Site 2306), São Paulo
- Princess Margaret Cancer Centre-Division of Medical Oncology and Hematology ( Site 0200), Toronto, Ontario, Canada
- Chile (7):
  - IC La Serena Research ( Site 2405), La Serena, Coquimbo Region
  - Oncocentro Valdivia ( Site 2407), Valdivia, Los Ríos Region
  - FALP-UIDO ( Site 2400), Santiago, Region M. de Santiago
  - Clínica Inmunocel ( Site 2404), Santiago, Region M. de Santiago
  - Clínica RedSalud Vitacura ( Site 2409), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 2403), Santiago, Region M. de Santiago
  - Biocenter ( Site 2401), Concepción, Región del Biobío
- China (16):
  - Beijing Cancer hospital ( Site 3000), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital-Medical Oncology ( Site 3025), Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital ( Site 3026), Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center-Internal Medicine ( Site 3001), Guangzhou, Guangdong
  - Zhujiang Hospital ( Site 3002), Guangzhou, Guangdong
  - The First Affiliated Hospital of Henan University of Science &Technology ( Site 3029), Luoyang, Henan
  - Henan Cancer Hospital-hematology department ( Site 3013), Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 3017), Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University ( Site 3004), Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital ( Site 3005), Nanchang, Jiangxi
  - The First Hospital of Jilin University-Hematology ( Site 3012), Changchun, Jilin
  - Fudan University Shanghai Cancer Center ( Site 3009), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University-Head and Neck Oncology ( Site 3016), Chengdu, Sichuan
  - Sichuan Cancer hospital-Oncology ( Site 3021), Chengdu, Sichuan
  - Zhejiang Cancer Hospital ( Site 3014), Hangzhou, Zhejiang
  - The First Affiliated Hospital Zhejiang University School of Medicine ( Site 3027), Hangzhou, Zhejiang
- Colombia (5):
  - Hospital Pablo Tobon Uribe ( Site 0804), Medellín, Antioquia
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 0801), Bogotá, Bogota D.C.
  - Instituto Médico de Alta Tecnologia S.A.S ( Site 0803), Montería, Departamento de Córdoba
  - Oncologos del Occidente ( Site 0800), Pereira, Risaralda Department
  - Fundacion Valle del Lili ( Site 0802), Cali, Valle del Cauca Department
- Costa Rica (2):
  - Hospital Metropolitano - Sede Lindora ( Site 2500), Santa Ana, Provincia de San José
  - CIMCA ( Site 2501), San José
- France (2):
  - centre hospitalier lyon sud-Service Hématologie ( Site 0702), Pierre-Bénite, Rhone
  - Pitie Salpetriere University Hospital-Clinical haematology ( Site 0700), Paris
- Greece (3):
  - Evangelismos General Hospital of Athens ( Site 0900), Athens, Attica
  - Regional General Hospital of Athens "Laiko" ( Site 0901), Athens, Attica
  - University Hospital of Alexandroupolis ( Site 0903), Alexandroupoli, East Macedonia and Thrace
- Guatemala (3):
  - MEDI-K ( Site 2602), Guatemala City
  - Private Practice- Dr. Rixci Augusto Lenin Ramírez ( Site 2601), Guatemala City
  - CELAN,S.A ( Site 2603), Guatemala City
- Hong Kong (2):
  - Queen Mary Hospital ( Site 3100), Hong Kong
  - Princess Margaret Hospital ( Site 3101), Hong Kong
- Israel (3):
  - Emek Medical Center-Hematology Unit ( Site 1102), Afula
  - Carmel Hospital ( Site 1103), Haifa
  - Hadassah Medical Center ( Site 1100), Jerusalem
- Italy (4):
  - Humanitas-U.O di Oncologia medica ed Ematologia ( Site 1203), Rozzano, Milano
  - IRCCS - AOU di Bologna-Istituto di Ematologia "L. e A. Seragnoli" ( Site 1200), Bologna
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 1202), Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -ISTITUTO DI EMATOLOGIA ( Site 1204), Roma
- Mexico (3):
  - Health Pharma Professional Research S.A. de C.V: ( Site 2700), Mexico City, Mexico City
  - Medivest Centro de Investigación Integral ( Site 2704), Chihuahua City
  - Centro de Infusion Superare ( Site 2701), Mexico City
- Aotearoa Clinical Trials ( Site 0501), Auckland, New Zealand
- Peru (4):
  - Clínicas AUNA Sede Chiclayo ( Site 2803), Chiclayo, Lambayeque
  - Clínica San Felipe ( Site 2805), Lima
  - Hospital Nacional Edgardo Rebagliati Martins ( Site 2802), Lima
  - Hospital Nacional Dos De Mayo ( Site 2804), Lima
- Poland (8):
  - Pratia MCM Krakow ( Site 1303), Krakow, Lesser Poland Voivodeship
  - Specjalistyczny Szpital im. Dr Alfreda Sokolowskiego w Walbrzychu ( Site 1305), Wałbrzych, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny-Klinika Hematologii, Nowotworow Krwi i Transplantacji Szpiku ( Site 1301), Wroclaw, Lower Silesian Voivodeship
  - Centrum Onkologii Ziemi Lubelskiej-Oddzial Hematologii i Transplantacji Szpiku ( Site 1304), Lublin, Lublin Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Układu Chłonnego ( Site 1300), Warsaw, Masovian Voivodeship
  - Szpitale Pomorskie Sp. z o. o.-Hematology and Bone Marrow Transplantation Department ( Site 1302), Gdynia, Pomeranian Voivodeship
  - Wojewódzki Szpital Specjalistyczny im. J. Korczaka w Słupsku ( Site 1309), Słupsk, Pomeranian Voivodeship
  - Pratia Onkologia Katowice ( Site 1306), Katowice, Silesian Voivodeship
- South Korea (2):
  - Seoul National University Hospital-Oncology ( Site 0302), Seoul
  - Samsung Medical Center ( Site 0300), Seoul
- Thailand (3):
  - Faculty of Medicine Siriraj Hospital-Division of Hematology, Department of Medicine ( Site 0400), Bangkok, Bangkok
  - Chulalongkorn University ( Site 0402), Pathumwan, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital ( Site 0401), Chiang Mai
- Turkey (Türkiye) (6):
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi ( Site 1912), Yenimahalle, Ankara
  - Ege University Medicine of Faculty ( Site 1902), Bornova, İzmir
  - Ankara University Hospital Cebeci-hematology ( Site 1901), Ankara
  - Mega Medipol-Hematology ( Site 1909), Istanbul
  - Dokuz Eylül Üniversitesi-Hematology ( Site 1905), Izmir
  - Ondokuz Mayıs Universitesi ( Site 1907), Samsun
- Ukraine (5):
  - MNPE ClinCenter of Oncology,Hematology,Transplantology and Palliative Care of CherkasyRegCouncil ( Site 2000), Cherkasy, Cherkasy Oblast
  - Communal non-profit enterprise "Regional clinical hospital of Ivano-Frankivsk Regional Council" ( Site 2004), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Institute of Blood Pathology and Transfusion Medicine AMS Ukraine ( Site 2002), Lviv, Lviv Oblast
  - State non-profit enterprise National Cancer Institute ( Site 2001), Kyiv
  - National Research Center for Radiation Medicine of National Academy of Medical Sciences of Ukraine ( Site 2005), Kyiv
- United Kingdom (3):
  - Aberdeen Royal Infirmary ( Site 2104), Aberdeen, Aberdeen City
  - The Royal Cornwall Hospital ( Site 2103), Truro, England
  - University College London Hospital-Cancer Clinical Trials Unit ( Site 2100), London-Camden, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26287&tenant=MT_MSD_9011